CLINICAL TRIAL: NCT00962234
Title: Metabolism of Lipids in Advanced Cancer
Status: Terminated | Type: Observational
Why Stopped: ethics approval not renewed by Study Group
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CIHR PIN 111846/ethics 24906; CIHR PIN 111846
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Lung Neoplasms; Cachexia
Keywords: Lipogenesis; Lipolysis; Phospholipids; Body Composition; Nutritional Status; Lipid Metabolism
MeSH Terms: conditions — Lung Neoplasms; Cachexia | interventions — Blood Specimen Collection; Deuterium; Deuterium Oxide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metabolism: Lung cancer patients who exhibit abnormalities in lipid measures.
  Interventions: Other: Blood draws; Biological: Oral administration of stable isotope (deuterium); Procedure: Metabolic rate testing

INTERVENTIONS:
Other: Blood draws — Up to 4 blood draws will be required, in the amount of about 10 mL each
Biological: Oral administration of stable isotope (deuterium) — 1 mg deuterium-labeled water/kg body water (loading dose), and 0.5 mg/kg body water diluted in 1 L of normal water (maintenance dose) to be consumed over the following 16 hours
  Other Names: C/D/N Isotopes, Deuterium Oxide, CAS No: 7789-20-0
Procedure: Metabolic rate testing — Metabolic rate testing is a painless, non-invasive test that takes about 1h. A metabolic cart is used, which detects the amount of oxygen and carbon dioxide the body uses. Patients will lie down on a bed for 30 minutes with lights dimmed and soft music to help them relax. After 30 minutes, a canopy will be placed over the patient's head and shoulders for 30 minutes for the analysis of breath samples. This test will be performed only once for this study.

SUMMARY:
The causes of failing nutrition status in advanced cancer are not well known. The way fat is moved, stored, burned or changed into other compounds may be affected and will be followed in patients using a tracer and other blood tests. The investigators hypothesize that fat loss and wasting results from low essential fatty acid availability in the body. Changes may occur in the liver that limits distribution and availability of fat to the body as an energy source or for other essential functions.

DETAILED DESCRIPTION:
Weight loss in cancer is the result of breakdown of fat (lipid) and muscle protein reserves. This research will explore how people with cancer use fat in their body through the use of tracers and measures in the blood. A stable isotope of hydrogen called 'deuterium' is used to trace the production of different fats by the liver. Other methods will determine how much and what types of fat are transported around the body. Body composition will be determined by CT scan and related to fat measures.

ELIGIBILITY:
Inclusion Criteria:

* Low plasma phospholipids OR low plasma ratio of triglycerides to free fatty acids
* Recent weight loss
* Advanced stage lung cancer (Stage 3 or 4)

Exclusion Criteria:

* Having symptoms that may affect measures of fat metabolism (nausea, vomiting, problems swallowing, etc.)
* Taking n-3 fatty acid supplements such as fish oil

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of hepatic de novo lipogenesis | 9 months

SECONDARY OUTCOMES:
Measures of fat transport and availability | 9 months
Resting metabolic rate & fat oxidation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Vera Mazurak, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada